CLINICAL TRIAL: NCT02528201
Title: A Twelve Week, Randomized, Double Blind Parallel Group Study Of Two Doses Of Celecoxib Compared To Diclofenac In Patients With Ankylosing Spondylitis
Brief Title: A Study Of Celecoxib Versus Diclofenac In Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COXA-0508-247; A3191099 (Other: Alias Study Number)
Record Dates: First submitted 2015-06-18; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Celecoxib; Diclofenac
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Celecoxib 200 milligrams mg QD (Active Comparator): celecoxib 200 milligrams (mg) once a day (QD)
  Interventions: Drug: Celecoxib 200 milligrams
- Celexocib 400 mg QD (Active Comparator): celecoxib 400 milligrams (mg) once a day (QD)
  Interventions: Drug: Celecoxib 400 milligrams
- Diclofenac 50 mg TID (Active Comparator): diclofenac 50 milligrams (mg) three times a day (TID)
  Interventions: Drug: diclofenac 50 milligrams

INTERVENTIONS:
Drug: Celecoxib 200 milligrams — Celecoxib 200 milligrams once a day
  Arms: Celecoxib 200 milligrams mg QD
Drug: Celecoxib 400 milligrams — Celecoxib 400 milligrams once a day
  Arms: Celexocib 400 mg QD
Drug: diclofenac 50 milligrams — diclofenac 50 milligrams three times a day
  Arms: Diclofenac 50 mg TID

SUMMARY:
A clinical trial to assess the effect of celecoxib 200 milligrams (mg) once daily and 400 milligrams (mg) once daily compared to diclofenac three times daily in the treatment of Ankylosing Spondylitis (AS) for 12 weeks. This will be used to confirm the results of a prior 6 week trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age, inclusive.
* Clinical diagnosis of ankylosing spondylitis:
* Willing to stop existing NSAID/COX-2 inhibitor treatment for up to two weeks.
* Having given written informed consent to participate in the trial.
* Pain intensity ≥ 40 mm on the visual analog scale, worsening by at least 30 % compared to that recorded at the screening visit.
* Last administration of analgesic without anti-inflammatory activity is ≥ 8 h, the last administration of long-acting NSAIDs is ≥ 72 h

Exclusion Criteria:

* Patients with acute peripheral articular disease (defined by the onset within 4 weeks prior to visit
* Known inflammatory enteropathy (e.g. ulcerative colitis, Crohn's disease).
* Ongoing extra-articular signs (e.g. cardiac involvement).
* Current painful vertebral compression.
* Requirement to start physiotherapy, re-education or manipulation
* History of clinical gastroduodenal ulcer in the year preceding inclusion, confirmed by endoscopy; continuing gastro-intestinal bleeding.
* Cardiac failure or known renal insufficiency that could be affected by study medication, chronic or acute hepatic insufficiency, significant coagulation disorders or history of asthma.
* Current or history of malignancy (except: patients having a basal cell carcinoma or other malignancy operated on and in remission for 5 years before inclusion in the trial).
* Pregnancy, women of childbearing potential not using adequate contraceptive methods or nursing mothers.
* Subject who has evidence of alcohol or drug abuse.
* Participation in any other clinical study within 30 days prior to the screening visit.
* Any condition that would prevent the patient from entering the study, according to the investigator's judgment.
* Known hypersensitivity to celecoxib, sulphonamides or any NSAID (including salicylic acid).
* Taking the following medications: Muscle relaxants, hypnotic, anxiolytics, sedatives, tranquillizers or antidepressants (unless stable for 2 weeks before screening and continuing throughout the trial), NSAIDs or COX-2 inhibitors other than study medication, acetylsalicylic acid (ASA) > 160 mg /day, anti-coagulants, ticlopidine, lithium, anti-TNF agents or methotrexate > 15 mg/week (Note: ASA ≤ 160 mg/day for cardioprotection is permitted), Use of oral or systemic analgesic medication, except from paracetamol, within 3 days of study entry and through the study, Corticosteroids (PO/IM/IV/IA) in the 6 weeks preceding inclusion in the trial, Anti-ulcer medication including chronic (daily or almost daily) use of antacids [Note: Occasional use of antacids during the study will be permitted.]
* Change in dose of a slow-acting drug (e.g. sulfasalazin, methotrexate) in the past 60 days preceding inclusion in the trial.
* Taking paracetamol > 2000 mg/day (including during the screening period).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2002-09; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Change in baseline of Patient Global Assessment of Pain Intensity (VAS) at week 12 | Baseline, Week 12
  Global Pain Intensity score (VAS): is a participant reported assessment of pain on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS) where 0 mm= no pain and 100=most severe pain.

SECONDARY OUTCOMES:
Participants Global Assessment of Pain Intensity (VAS) | Weeks 2, 6
  Global Pain Intensity score (VAS): is a participant reported assessment of pain on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS) where 0 mm= no pain and 100=most severe pain.
Bath Ankylosing Spondylitis Functional Index (BASFI) | Weeks 2, 6
  BASFI is a validated self assessment tool that determines the degree of functional limitation in AS. Utilizing a VAS of 0-10 (0 = easy, 10 = impossible), participants answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a mean score of the 10 questions.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Weeks 2, 6
  BASDAI is a validated self assessment tool used to determine disease activity in participant with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The final BASDAI score averages the individual assessments for a final score range of 0-10
Participants and Physicians Global Assessment of Disease Activity | Weeks 2, 6, 12
  Participants are asked at each visit the following questions: Taking everything into account how do you assess the activity of your disease in the last 2 days on a scale where: 0=disease inactive with no symptoms and 100=disease extremely active?
Participants and Physicians Global Assessment of Treatment | Week 12
  The patients will be asked up to four global questions about safety and efficacy of the trial medication and about their current disease status. Responses are done on a 5 point scale where 0=no effect, 1=poor effect, 2=moderate effect, 3=good effect, and 4=excellent. At the same visits the investigator will be asked to do his/her own judgment of the efficacy and tolerance of the treatment (excellent, good, moderate, poor).
Participants Consumption of Rescue Medication | Baseline, Weeks 2, 6, 12
  Participant consumption of rescue medication (paracetamol) calculated at each individual visit (except from the screening visit) by counting returned tablets versus tablets dispensed at the previous visit.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Norway (27):
  - Ålesund sykehus, Ålesund
  - Bekkestua legesenter, Bekkestua
  - Dr. Johannessen Kontor, Bergen
  - Dr.Wiigs kontor, Bergen
  - Nordland Medisinske Senter, Bodø
  - Martina Hansens hospital, Bærum Postterminal
  - Sykehuset Buskerud HF, Drammen
  - Lægene på Kongens torv, Gamle Fredrikstad
  - Centre For Clinical Trials, Hamar
  - Harstad sykehus, Harstad
  - Haugesund sanitetsforenings revmatismesykehus, Haugesund
  - Horten legesenter, Horten
  - Solli Klinikk AS, Jessheim
  - Kongsvinger sykehus HF, Kongsvinger
  - Vest-Agder sentralsykehus, Kristiansand
  - Dr. Svensens kontor, Kristiansand
  - Lensbygda Legekontor, Lena
  - Helse Nord-Trøndelag HF, Sykehuset Levanger, Levanger
  - LSF Reumatismesykehus, Lillehammer
  - Helgelandssykehuset HF, Mo i Rana
  - Rikshospitalet, Oslo
  - Økernlegene, Oslo
  - Diakonhjemmet Hospital, Oslo
  - Betanien Hospital, Skien
  - Rosten legesenter, Tiller
  - Universitetssykehuset Nord-Norge HF, Tromsø
  - St.Olavs Hospital, Trondheim